CLINICAL TRIAL: NCT06834750
Title: The Application of Kinesio Taping Technique in the Early Upper Limb Functional Activities Induction of Hemiplegic Patients After Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2024-244
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Infarction Recovery; Rehabilitation Treatment; Upper Extremity Motor Function; Emg Biofeedback
Keywords: Ischemia; Necrosis; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Stroke; Vascular Diseases; Cardiovascular Diseases; Cerebral Infarction; Infarction
MeSH Terms: conditions — Ischemia; Necrosis; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Stroke; Vascular Diseases; Cardiovascular Diseases; Cerebral Infarction; Infarction | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): The control group was pasted with sports white tape.
  Interventions: Other: Control group (placebo)
- experimental group (Experimental): The experimental group received intramuscular patch therapy.
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Experimental Group — The application methods of kinesiology tape for the experimental group are as follows:
  1. Promoting supraspinatus muscle: Use an I-shaped tape (with natural tension).
  2. Promoting the anterior fibers of the deltoid muscle: Use an I-shaped tape (with natural tension).
  3. Promoting the posterior fibers of the deltoid muscle: Use an I-shaped tape (with natural tension).3. Promoting the posterior fibers of the deltoid muscle: Use an I-shaped tape (with natural tension).
  4. Fixing the shoulder joint: Use an I-shaped tape (with moderate tension).
  5. Inhibiting biceps brachii muscle / promoting triceps brachii muscle (depending on the patient's recovery stage and different functional impairments, different taping methods are used).
  6. Promoting wrist extensor muscles / inhibiting wrist flexor muscles (depending on the patient's recovery stage and different functional impairments, different taping methods are used)
  Arms: experimental group
Other: Control group (placebo) — The control group was pasted with sports white tape (the pasting method was the same as above, replaced with sports white tape).
  Arms: control group

SUMMARY:
1. To observe the inducing and promoting effect of kinesio taping technique on the recovery of upper limb function in early-stage stroke patients.
2. To compare the different effects of kinesio tape and sports white tape on the induction and promotion of limb function in patients.
3. To verify that kinesio taping technique is a safe and promotable technical means for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the experiment and signed informed consent
2. Diagnosed as a stroke patient
3. No other major cardiovascular and cerebrovascular diseases
4. First new stroke
5. After evaluation by evaluators, subjects had Brunnstrom stage < 3

Exclusion Criteria:

1. The subject's compliance was poor
2. Increased muscle tone in the affected upper extremity
3. Subjects with skin allergies
4. Those who did not receive continuous treatment during the experiment

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
To observe the inducing and promoting effect of kinesio taping technique on the recovery of upper limb function in early-stage stroke patients. | Within 3 days of hospitalization, on the 1 day of discharge, one month after discharge
  Fugl-Meyer Functional Score (FMA) is evaluated, and the higher the score, the stronger the motor function.

SECONDARY OUTCOMES:
To compare the different effects of kinesio tape and sports white tape on the induction and promotion of limb function in patients. | Within 3 days of hospitalization, on the 1 day of discharge, one month after discharge
  Fugl-Meyer Functional Score (FMA) is evaluated, and the higher the score, the stronger the motor function.

CONTACTS AND LOCATIONS:
Locations (1):
- 4th Affiliated Hospital, School of Medicine, Zhejiang University, China, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No